CLINICAL TRIAL: NCT02472236
Title: An Open-label,Sequential,Single-site Study to Evaluate the Pharmacokinetics of Digoxin When Coadministered With Polyethylene Glycol Loxenatide (PEX168) in Healthy Adult Subjects
Brief Title: Evaluate the Pharmacokinetics of Digoxin When Coadministered With PEX168 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PEX168-Ij
Record Dates: First submitted 2015-05-26; First posted 2015-06-15 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2016-01

CONDITIONS: Healthy
Keywords: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — polyethylene glycol loxenatide; Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Digoxin and PEX168(200µg) (Experimental): Digoxin: 0.5mg, oral Administration. PEX 168: 200µg,injected subcutaneously,once a week.
  Interventions: Drug: PEX168; Drug: Digoxin

INTERVENTIONS:
Drug: PEX168 — 200µg,injected subcutaneously,once a week.
  Other Names: Polyethylene Glycol Loxenatide
Drug: Digoxin — 0.5mg,oral,two times.
  Other Names: Digaoxin tablet

SUMMARY:
To assess the effect of PEX168 doses on the pharmacokinetics of digoxin in healthy subjects.To provide a scientific basis for clinical drug combination of PEX168.

To assess the safety of single doses of digoxin administered with and without PEX168

DETAILED DESCRIPTION:
This was an open-label, sequential, single-center study that evaluated the pharmacokinetics of digoxin when coadministered with PEX168 in healthy adult subjects. The total duration of each subject's participation in the study was approximately 12 weeks, which included up to a 14-day Screening Period, a 44-day Treatment Period, and an approximately 4-week Follow-up Period.

Center: This study was conducted at a single site in the first affiliate hospital of Xi'an Jiaotong University.All subjects receives a single 0.5mg oral dose of digoxin on Day 1 followed by 5 weekly 200μg doses of PEX168 injected subcutaneously beginning on Day 8 and a second single 0.5mg oral dose of digoxin on Day 38.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male aged 18 to 45 years (including both ends) at the time of signing the informed consent.
2. Weighing not less than 50kg，Body Mass Index (BMI)of 18 to 25kg/m2.
3. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), total bilirubin (Tbil) are within the normal range during screening;
4. Estimated creatinine clearance (Clcr) ≥90ml / min calculated by the Cockcroft-Gault (CG) formula ;
5. Capable of giving written informed consent, which included compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

1. The hepatitis B surface antigen, hepatitis C antibody, HIV antibody test positive;
2. Having history of syncope, palpitations, bradycardia, tachycardia and other anomalies(such as the extent of any way block, left bundle branch block, right bundle branch block), or via a comprehensive physical examination (vital signs, physical examination), routine laboratory tests (blood count, blood biochemistry, urine, etc.), 12-lead ECG, abdominal B ultrasound (liver, gallbladder, pancreas, spleen, kidney), and other abnormalities and clinical significance persons before screening;
3. Having Alcohol and drug abuse within first 6 months before screening;
4. Smoked within 3 months before screening;
5. In screening period, blood pressure greater than 140 / 90mmHg, retest after diagnosis or pulse rate is higher than 100bpm person;
6. In screening period, ECG QTc> 450ms,diagnosed after retest;
7. Having a history of drug or allergic reactions or allergic constitution have hypersensitivity to any of the following:

1) digoxin and / or any of its ingredients or other similar drugs . 2) PEX168

8. Before screening, having a history of cardiovascular disease (coronary heart disease, high blood pressure, high cholesterol, etc.) or a history of pulmonary disease (chronic bronchitis, emphysema, asthma, pneumonia, etc.);

9. In screening period , fasting triglycerides test result was greater than the upper limit of normal range;

10. Currently there is a history of liver disease or liver disease or a known hepatobiliary abnormalities (except asymptomatic gallstones);

11. Participate in blood donation and donation amount ≥400ml within three months before screening, or who participate in blood donation or blood transfusion within a month;

12. In screening period, having thyroid dysfunction or a history;

13. The history of gastrointestinal surgery (such as stomach cutting surgery, gastric bypass surgery) before screening;

14. The history of pancreatitis;

15. History of cholecystitis gallbladder disease or other disease history;

16. The history of inflammatory bowel disease or a history of irritable bowel syndrome;

17. The history of Type 2 multiple endocrine neoplasia;

18. The history of medullary thyroid cancer;

19. The family has type 2 multiple endocrine fibromatosis or a history of medullary thyroid cancer;

20. 3 months before screening, participating in any drug or medical device trials are (including placebo);

21. Using any of the tested drugs may affect prescription drugs , non-prescription drugs, herbal (especially ginseng, oral hypoglycemic agents) or multivitamin supplements persons;

22. Drinking medication or caffeine-containing xanthine food and beverage (listed in annex 3), strenuous exercise, or other effects of drug absorption, distribution, metabolism, excretion and other factors 2 days before screening.

23. Received GLP-1 analogs (e.g. exenatide) treatment;

24. Reluctant to take an effective method of contraception during the test, fertility planner within six months after his or her spouse during the test or the last dose (38 days);

25. Researchers believe any situation that might lead to any subject cannot complete the study or to the subject of this study bring significant risk.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-06-08 (Actual); Primary Completion 2015-09-24 (Actual); Study Completion 2016-01-18 (Actual)

PRIMARY OUTCOMES:
Composite measure the plasma concentrations of Digoxin. | Baseline to Day44
  Plasma concentrations of digoxin, and to calculate the pharmacokinetic parameters: Tmax、Cmax、AUC0-t、AUC0-∞、λz ，t1/2、Vd/F、CLr etc.

SECONDARY OUTCOMES:
Incidence of adverse events and serious adverse events | Baseline to Day72

CONTACTS AND LOCATIONS:
Overall Officials: Bingyin Shi, Principal Investigator — The first affiliate of Xi'an Jiaotong University
Locations (1):
- The first affiliate of Xi'an Jiaotong University, Xi’an, Shanxi, China